CLINICAL TRIAL: NCT00578383
Title: Low Field Magnetic Stimulation in Mood Disorders Using the LFMS Device
Acronym: LFMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006-P-001655; Stanley Grant 07TGS-1045 (Other Grant/Funding Number: Stanley Grant 07TGS-1045)
Record Dates: First submitted 2007-12-18; First posted 2007-12-21 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Depression; Bipolar Depression; Major Depressive Disorder
Keywords: Depression; Major depression; Bipolar Disorder; Bipolar depression; LFMS; low field magnetic stimulation; mood disorders; affective disorders
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sham (inactive) Treatment BPD (Sham Comparator): 20 minutes of sham treatment with the Low Field Magnetic Stimulation Device (LFMS)in bipolar depressed subjects
  Interventions: Device: Low Field Magnetic Stimulation Device
- Active LFMS treatment in BPD (Active Comparator): 20 minutes of active treatment with the Low Field Magnetic Stimulation Device (LFMS)in bipolar depressed subjects
  Interventions: Device: Low Field Magnetic Stimulation Device
- Sham LFMS Comparator: in MD (Sham Comparator): 20 minutes of sham treatment with the Low Field Magnetic Stimulation Device (LFMS) in major depressed subjects
  Interventions: Device: Low Field Magnetic Stimulation Device
- Experimental LFMS: in MD (Active Comparator): 20 minutes of active treatment with the Low Field Magnetic Stimulation Device (LFMS) in major depressed subjects
  Interventions: Device: Low Field Magnetic Stimulation Device

INTERVENTIONS:
Device: Low Field Magnetic Stimulation Device — The LFMS Device is an electromagnetic coil situated on a cylinder with an inside diameter of 13.2 inches. It produces weak electromagnetic fields at a frequency of about 1 kHz; the magnetic fields are less than 30 Gauss and the electric fields are up to 1.43 V/m. Subjects will receive one 20 minute treatment.
  Other Names: LFMS

SUMMARY:
This study is designed to test whether low-field magnetic stimulation (LFMS) can relieve some of the symptoms of depression in bipolar disorder or major depression.

DETAILED DESCRIPTION:
This study involves a screening visit with the study physician and a treatment visit. Participants will be asked to complete several questionnaires about their mood during both visits. The treatment visit will involve use of the LFMS device. Participants will place the top of their head inside the device for approximately 20 minutes. Participants will receive either the actual treatment or a sham treatment and will not know which they receive. This device produces weak electromagnetic fields. There is no discomfort or even sensation caused by the device. The device has been declared to be a "non-significant risk device" by the FDA, and there are no known risks associated with its use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder or Bipolar Disorder; must be currently depressed
* May be medicated or unmedicated

Exclusion Criteria:

* Contraindication for MRI due to metal in eyes/head
* Claustrophobia.
* Inability to lie flat.
* History of brain injury.
* Pregnant
* Current drug use/abuse/dependence
* History of polysubstance use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-11; Primary Completion 2011-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rohan, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Carlezon WA Jr, Rohan ML, Mague SD, Meloni EG, Parsegian A, Cayetano K, Tomasiewicz HC, Rouse ED, Cohen BM, Renshaw PF. Antidepressant-like effects of cranial stimulation within a low-energy magnetic field in rats. Biol Psychiatry. 2005 Mar 15;57(6):571-6. doi: 10.1016/j.biopsych.2004.12.011. PMID 15780843
- [Background] Rohan M, Parow A, Stoll AL, Demopulos C, Friedman S, Dager S, Hennen J, Cohen BM, Renshaw PF. Low-field magnetic stimulation in bipolar depression using an MRI-based stimulator. Am J Psychiatry. 2004 Jan;161(1):93-8. doi: 10.1176/appi.ajp.161.1.93. PMID 14702256
- [Derived] Rohan ML, Yamamoto RT, Ravichandran CT, Cayetano KR, Morales OG, Olson DP, Vitaliano G, Paul SM, Cohen BM. Rapid mood-elevating effects of low field magnetic stimulation in depression. Biol Psychiatry. 2014 Aug 1;76(3):186-93. doi: 10.1016/j.biopsych.2013.10.024. Epub 2013 Nov 12. PMID 24331545
- See also: Link to McLean Hospital clinical study website — http://www.mclean.harvard.edu/research/clinical/study.php?sid=123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from March 2008 though February 2011. They were recruited through flyers distributed around McLean Hospital (Belmont, MA), referral by clinic doctors and direct recruitment on the hospital's units.
Pre-assignment Details: Enrolled participants are excluded from statistical results if they had baseline Hamilton Depression Rating scores under 17 or co-morbid disorders.
Groups:
- Bipolar Disorder Active LFMS Treatment: Subjects with bipolar depression receiving active treatment with the Low Field Magnetic Stimulation Device.
- Bipolar Disorder Sham LFMS Treatment: Subjects with bipolar depression receiving sham treatment with the Low Field Magnetic Stimulation Device. The sham treatment is identical to the active treatment, with the exception that subjects to not receive the active stimulation.
- Major Depressive Disorder Active LFMS Treatment: Subjects with major depression receiving active treatment with the Low Field Magnetic Stimulation Device.
- Major Depressive Disorder Sham LFMS Treatment: Subjects with major depression receiving sham treatment with the Low Field Magnetic Stimulation Device. The sham treatment is identical to the active treatment, with the exception that subjects to not receive the active stimulation.
Period: Overall Study
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Started | 37 | 36 | 19 | 15
Completed | 21 | 20 | 13 | 9
Not Completed | 16 | 16 | 6 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled participants are excluded from statistical results if they had baseline Hamilton Depression Rating scores under 17 or co-morbid disorders.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment | Total
Number analyzed (Participants) | 37 | 36 | 19 | 15 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 19 | 15 | 106
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.0) | 42.2 (12.2) | 43.1 (15.5) | 43.5 (14.9) | 42.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 15 | 12 | 8 | 60
  Male | 12 | 21 | 7 | 7 | 47
Region of Enrollment [Number; unit: participants]
  United States | 37 | 36 | 19 | 15 | 107

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change in Hamilton Depression Rating Scale (HAM-D) (17 Item): Combined Diagnostic Groups.
Description: A multiple choice questionnaire used to rate depression severity. Mean change from pretreatment score. 17 items reflecting depression symptoms are scored on scale of severity; 9 items are scored 0 = Absent 1 = Trivial 2 = Mild 3 = Moderate 4 = Severe 8 items are scored 0 = Absent 1 = Mild 2 = Severe. Items are summed; minimum score is 0, maximum score is 52. Higher scores represent more severe depression.
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Combined Group Active LFMS Treatment: Combined diagnostic groups receiving active treatment with the Low Field Magnetic Stimulation Device.
- Combined Group Sham LFMS Treatment: Combined diagnostic groups receiving sham treatment with the Low Field Magnetic Stimulation Device. The sham treatment is identical to the active treatment, with the exception that subjects to not receive the active stimulation.
Arm/Group | Combined Group Active LFMS Treatment | Combined Group Sham LFMS Treatment
Number analyzed (Participants) | 32 | 29
units on a scale | -8.13 (0.87) | -5.02 (0.78)
Statistical Analysis 1: Comparison: Combined Group Active LFMS Treatment vs Combined Group Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression and those with major depressive disorder as assessed by the 17-item Hamilton Depression Rating Scale; Test type: Superiority or Other; p = 0.009, Regression, Linear — We used type HC3 robust standard errors (SEs)in place of OLS regression SEs to guard against biased estimation of SEs due to heteroscedasticity. This is an uncorrected p-value with a required threshold of 0.025 for significance (correction factor 2); Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 3.11, 95% CI 2-sided [0.5 to 5.8], Standard Error of Mean 1.17

2. Secondary Outcome: Visual Analog Scale (VAS): Combined Diagnostic Groups.
Description: Eleven point Likert scales indicating immediate depression state. Mean change from pretreatment score. Participant marks an 'X' on a numbered line anchored by 0 = no depression and 10 = most depressed ever been.
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Combined Groups Sham LFMS Treatment: Combined diagnostic groups receiving sham treatment with the Low Field Magnetic Stimulation Device. The sham treatment is identical to the active treatment, with the exception that subjects to not receive the active stimulation.
Arm/Group | Combined Group Active LFMS Treatment | Combined Groups Sham LFMS Treatment
Number analyzed (Participants) | 34 | 29
units on a scale | -1.66 (0.29) | -0.60 (0.23)
Statistical Analysis 1: Comparison: Combined Group Active LFMS Treatment vs Combined Groups Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression and those with major depressive disorder as assessed by a visual analog scale; Test type: Superiority or Other; p = 0.006, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 1.06, 95% CI 2-sided [0.2 to 1.9], Standard Error of Mean 0.38

3. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Positive Score: Combined Diagnostic Group.
Description: 20 item list of words that describe different feelings and emotions with positive and negative valences (10 each), which the subject scores on a 1-5 scale: 1 = very slightly or not at all 2 = a little 3 = moderate 4 = quite a bit 5 = extremely. Positive and Negative scores are calculated and reported separately and range from 10-50. Higher positive score reflects stronger positive affect and higher negative score reflects stronger negative affect.
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Combined Groups Active LFMS Treatment: Combined diagnostic groups receiving active treatment with the Low Field Magnetic Stimulation Device.
Arm/Group | Combined Groups Active LFMS Treatment | Combined Groups Sham LFMS Treatment
Number analyzed (Participants) | 34 | 29
units on a scale | 3.16 (0.93) | -0.94 (0.79)
Statistical Analysis 1: Comparison: Combined Groups Active LFMS Treatment vs Combined Groups Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression and those with major depressive disorder as assessed by the PANAS (POSITIVE SCALE); Test type: Superiority or Other; p = 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 4.1, 95% CI 2-sided [1.3 to 6.9], Standard Error of Mean 1.24

4. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Negative Score: Combined Diagnostic Group.
Description: as for outcome 3
Time Frame: once pre and once post LFMS treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combined Groups Active LFMS Treatment | Combined Groups Sham LFMS Treatment
Number analyzed (Participants) | 34 | 29
units on a scale | -7.00 (1.02) | -5.00 (0.91)
Statistical Analysis 1: Comparison: Combined Groups Active LFMS Treatment vs Combined Groups Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression and those with major depressive disorder as assessed by the PANAS (negative scale); Test type: Superiority or Other; p = 0.15, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 2.0, 95% CI 2-sided [-1.1 to 5.1], Standard Error of Mean 1.39

5. Primary Outcome: Mean Change in Hamilton Depression Rating Scale (HAM-D) (17 Item) in Subjects With Bipolar Depression
Description: as for outcome 1
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment
Number analyzed (Participants) | 19 | 20
units on a scale | -8.3 (1.0) | -5.79 (1.07)
Statistical Analysis 1: Comparison: Bipolar Disorder Active LFMS Treatment vs Bipolar Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression as assessed by the 17-item Hamilton Depression Rating Scale; Test type: Superiority or Other; p = 0.09, Regression, Linear — We used type HC3 robust standard errors (SEs)in place of OLS regression SEs to guard against biased estimation of SEs due to heteroscedasticity. This is an uncorrected p-value with a required threshold of 0.0125 for significance (correction factor 4); Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 2.5, 95% CI 2-sided [-1.2 to 6.2], Standard Error of Mean 1.47

6. Primary Outcome: Mean Change in Hamilton Depression Depression Rating Scale (HAM-D) (17 Item) in Subjects With Major Depressive Disorder
Description: as for outcome 1
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Major Depressive Disorder Sham LFMS Treatment: Subjects with major depression receiving sham treatment with the Low Field Magnetic Stimulation Device. The sham treatment is identical to the active treatment, with the exception that subjects to not receive the active
Arm/Group | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Number analyzed (Participants) | 10 | 9
units on a scale | -7.19 (1.44) | -4.02 (1.54)
Statistical Analysis 1: Comparison: Major Depressive Disorder Active LFMS Treatment vs Major Depressive Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with major depressive disorder as assessed by the 17-item Hamilton Depression Rating Scale; Test type: Superiority or Other; p = 0.19, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 3.2, 95% CI 2-sided [-3.3 to 9.6], Standard Error of Mean 2.11

7. Primary Outcome: Visual Analog Scale (VAS) in Subjects With Bipolar Depression
Description: as for outcome 2
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment
Number analyzed (Participants) | 21 | 20
units on a scale | -1.18 (0.37) | -1.05 (0.35)
Statistical Analysis 1: Comparison: Bipolar Disorder Active LFMS Treatment vs Bipolar Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression as assessed by a visual analog scale; Test type: Superiority or Other; p = 0.15, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 0.76, 95% CI 2-sided [-0.6 to 2.1], Standard Error of Mean 0.51

8. Primary Outcome: Visual Analog Scale (VAS) in Subjects With Major Depressive Disorder
Description: as for outcome 2
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Number analyzed (Participants) | 13 | 9
units on a scale | -1.33 (0.53) | 0.25 (0.25)
Statistical Analysis 1: Comparison: Major Depressive Disorder Active LFMS Treatment vs Major Depressive Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with major depressive disorder as assessed by a visual analog scale; Test type: Superiority or Other; p = 0.04, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 1.58, 95% CI 2-sided [-0.4 to 3.6], Standard Error of Mean 0.67

9. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Positive Score in Subjects With Bipolar Depression.
Description: as for outcome 3
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment
Number analyzed (Participants) | 21 | 20
units on a scale | 4.18 (1.37) | -0.79 (0.93)
Statistical Analysis 1: Comparison: Bipolar Disorder Active LFMS Treatment vs Bipolar Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression as assessed by the PANAS (positive scale); Test type: Superiority or Other; p = 0.004, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 5.0, 95% CI 2-sided [0.8 to 9.2], Standard Error of Mean 1.67

10. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Positive Score in Subjects With Major Depressive Disorder
Description: as for outcome 3
Time Frame: Once just before and once just after treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Number analyzed (Participants) | 13 | 9
units on a scale | 1.05 (1.07) | -0.63 (1.11)
Statistical Analysis 1: Comparison: Major Depressive Disorder Active LFMS Treatment vs Major Depressive Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with major depressive disorder as assessed by the PANAS (positive scale); Test type: Superiority or Other; p = 0.30, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 1.7, 95% CI 2-sided [1.3 to 5.8], Standard Error of Mean 1.58

11. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Negative Score in Subjects With Bipolar Depression
Description: as for outcome 3
Time Frame: once pre and once post LFMS treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment
Number analyzed (Participants) | 21 | 20
units on a scale | -7.66 (1.45) | -6.31 (1.39)
Statistical Analysis 1: Comparison: Bipolar Disorder Active LFMS Treatment vs Bipolar Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with bipolar depression as assessed by the PANAS (negative scale); Test type: Superiority or Other; p = 0.52, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 1.3, 95% CI 2-sided [-4.1 to 6.8], Standard Error of Mean 2.01

12. Secondary Outcome: Positive and Negative Affect Schedule (PANAS) Negative Score in Subjects With Major Depressive Disorder
Description: as for outcome 3
Time Frame: once pre and once post LFMS treatment
Population: Qualifying subjects who completed the the study with qualifying HAM-D scores and complete data.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Number analyzed (Participants) | 13 | 9
units on a scale | -5.28 (1.10) | -3.04 (0.63)
Statistical Analysis 1: Comparison: Major Depressive Disorder Active LFMS Treatment vs Major Depressive Disorder Sham LFMS Treatment; Active LFMS treatment would reduce depression immediately after treatment in subjects with major depressive disorder as assessed by the PANAS (negative scale); Test type: Superiority or Other; p = 0.10, Regression, Linear — [p-value comment as in outcome 5, analysis 1]; Bonferroni multiple testing corrections were applied separately to results for our primary and secondary outcomes; Mean Difference (Net) = 2.2, 95% CI [-1.3 to 5.8], Standard Error of Mean 1.43

ADVERSE EVENTS:
Time Frame: 2 years, 10 months
Description: participant self report
Arm/Group | Bipolar Disorder Active LFMS Treatment | Bipolar Disorder Sham LFMS Treatment | Major Depressive Disorder Active LFMS Treatment | Major Depressive Disorder Sham LFMS Treatment
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/37 | 2/36 | 0/19 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Disorder Active LFMS Treatment (N=37) | Bipolar Disorder Sham LFMS Treatment (N=36) | Major Depressive Disorder Active LFMS Treatment (N=19) | Major Depressive Disorder Sham LFMS Treatment (N=15)
dizziness at venepuncture (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — dizziness at the sight of blood - psychological

LIMITATIONS AND CAVEATS:
A limitation of the current trial was that it was underpowered to detect moderate but clinically significant benefits of LFMS in diagnostic subgroups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No